CLINICAL TRIAL: NCT00282412
Title: Rheumatoid Arthritis: Tolerance Induction by Mixed Chimerism
Brief Title: Rheumatoid Arthritis:Tolerance Induction by Mixed Chimerism
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: No participant enrolled for three years. No plan to continue study.
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Richard Burt, MD, MD, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DIAD RA ALLO
Record Dates: First submitted 2006-01-24; First posted 2006-01-26 (Estimated); Results first posted 2018-07-30 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2017-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Hematopoietic Stem Cell Transplantation; fludarabine; fludarabine phosphate; Cyclophosphamide; Alemtuzumab; Filgrastim; Cyclosporins; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hematopoietic Stem Cell Transplantation (Experimental): Allogeneic Hematopoietic Stem Cell Transplantation will be performed on eligible patients diagnosed with RA
  Interventions: Biological: Hematopoietic Stem Cell Transplantation; Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Campath 1H; Drug: GCSF; Drug: Cyclosporins; Drug: Mycophenolate Mofetil

INTERVENTIONS:
Biological: Hematopoietic Stem Cell Transplantation — Allogeneic Hematopoietic Stem Cell Transplantation
Drug: Fludarabine — inhibits DNA synthesis or repair
  Other Names: Fludara
Drug: Cyclophosphamide — Causes prevention of cell division by forming adducts with DNA
  Other Names: Cytoxan, Neosar
Drug: Campath 1H — humanized monoclonal antibody against CD52 antigen
  Other Names: Alemtuzumab
Drug: GCSF — Hematopoietic growth factor
  Other Names: Neupogen
Drug: Cyclosporins — immune suppressive drug
  Other Names: CSA
Drug: Mycophenolate Mofetil — immune suppressive drug
  Other Names: Cellcept

SUMMARY:
Rheumatoid arthritis disease is believed to be due to immune cells, cells that normally protect the body and are now causing damage to the body. Risk of death is highest in people with twenty or more joints actively involved with disease, positive rheumatoid factor, an elevated sedimentation rate (laboratory measures of active inflammation), and patients with limitation of daily activities (trouble doing simple things like opening a carton of milk). In these high risk patients, life is significantly shortened. Death is usually from heart disease, kidney failure, neck dislocation, broken hip bones, or blood clots to the lung. In this study we use moderate dose chemotherapy (cyclophosphamide and fludarabine) and CAMPATH-1H (a protein that kills the immune cells that are thought to be causing the disease), followed by infusion of blood stem cells that have been collected from the patient's brother or sister (allogeneic stem cell transplant). The purpose of the moderate dose chemotherapy and CAMPATH-1H is to destroy the cells in the immune system and to allow the cells from the patient's brother or sister to grow. The purpose of the stem cell infusion is to restore blood cell production, which will be severely impaired by the moderate dose chemotherapy and CAMPATH-1H, and to produce a normal immune system that will no longer attack the body.

DETAILED DESCRIPTION:
Peripheral blood stem cell mobilization (PBSC)

PBSC will be mobilized with G-CSF (dose may be adjusted down to 5-10 ug/kg/day by PI for toxicity, e.g. flu-like symptoms) with stem cell collection beginning on day 4 or 5. Leukapheresis may be repeated up to four consecutive days.

Conditioning Regimen Immune Ablation:

Fludarabine 25 mg/m2/d x 5 days (dosage should be based on adjusted body weight) will be given IV over 30 minutes in 100 cc of normal saline.

Cyclophosphamide 50 mg/kg/d x 4 days (dosage should be based on adjusted body weight) will be given IV over 1 hour in 500 cc of normal saline.

CAMPATH-1H 30 mg/day x 3 days (no dose adjustment) will be given IV over 2 hours in 100 cc of normal saline. Premedication with acetaminophen 650mg & benadryl 25-50mg PO/IV will be given 30-60min before infusion. These medications can be repeated as needed.

Hydration approximately 200 cc /hour beginning 6 hours before cyclophosphamide and continued until 24 hours after the last cyclophosphamide dose.

G-CSF will be continued until absolute neutrophil count reaches 1,000 cells/ml for three days.

Cyclosporine will be started at 200 mg po BID and adjusted by HPLC levels to between 150-250 or by toxicity (e.g. tremor, renal insufficiency, TTP, etc.). CSA will be continued for 6 months unless stopped for toxicity

Mycophenolate Mofetil (Cellcept) will be given 1 gram po BID and may be adjusted by toxicity (e.g. cytopenia). Cellcept will be continued for 6 months unless stopped for toxicity.

ELIGIBILITY:
Participant Inclusion Criteria:

* Age > 18 and < 60 years at time of pre-transplant evaluation.
* An established clinical diagnosis of rheumatoid arthritis by American College of Rheumatology criteria.
* Patients must have failed an autologous hematopoietic transplant or have failed to respond to either methotrexate or leflunomide in combination with a TNF inhibitor. Failure is defined as an inability to tolerate treatment with at least 6 swollen joints and 20 involved joints or inability to answer at least 70% of HAQ questions with "no difficulty" despite 2 or more months of treatment.

  * Ability to give informed consent.
  * Patient must have a HLA matched sibling donor at the A, B, C, and DR loci to proceed or HLA matched cord blood donor.
  * If donor is HLA matched cord blood, cord blood stem cells will be obtained from the NMDP (1-800-548-1375) and one or two units of HLA matched cord blood will be infused on day zero.

Participant Exclusion Criteria

* History of coronary artery disease, or documented congestive heart failure.
* HIV positive.
* Uncontrolled diabetes mellitus, or any other illness that in the opinion of the investigators would jeopardize the ability of the patient to tolerate aggressive chemoradiotherapy.
* Prior history of malignancy except localized basal cell or squamous skin cancer. Other malignancies for which the patient is judged to be cured by local surgical therapy, such as head and neck cancer, or stage I breast cancer will be considered on an individual basis.
* Positive pregnancy test, inability or unwillingness to pursue effective means of birth control, failure to willingly accept or comprehend irreversible sterility as a side effect of therapy.
* Psychiatric illness or mental deficiency making compliance with treatment or informed consent impossible.
* FEV1/FVC < 70% of predicted, DLCO < 40% of predicted.
* Resting LVEF < 45 %.
* Bilirubin > 2.0 mg/dl (unless due to Gilberts), transferase (AST) > 2.5 x upper limit of normal.
* Serum creatinine > 2.0 mg/dl.

Donor Exclusion Criteria

* Age < 18 years.
* Positive for HIV-1, HIV-2, HTLV-I, HTLV-II.
* Active hepatitis B or C.
* History of a malignancy except for a localized cancer such as skin cancer that is deemed cured.
* History of myocardial infarction or congestive heart failure.
* Inability to give informed consent.
* Current pregnancy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2002-09; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Burt, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Feinberg School of Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hematopoietic Stem Cell Transplantation
Started | 4
Completed | 2 (Two late deaths non-treatment related. One from pulmonary embolism and one from late leukemia.)
Not Completed | 2
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Arm/Group | Hematopoietic Stem Cell Transplantation
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.00 (12.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Survival
Description: The number of participants who survived treatment
Time Frame: up to 5 years
Population: The number of participants who survived treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Hematopoietic Stem Cell Transplantation
Number analyzed (Participants) | 4
Participants | 2

ADVERSE EVENTS:
Time Frame: Up to 5 years
Description: All adverse events will be collected at 6 months, 1 year and then yearly up to five years
Arm/Group | Hematopoietic Stem Cell Transplantation
All-Cause Mortality (participants affected / at risk) | 2/4
Serious Adverse Events (participants affected / at risk) | 2/4
Other Adverse Events (participants affected / at risk) | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hematopoietic Stem Cell Transplantation (N=4)
Acute leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — One patient was in complete remission, RF neg, no GVHD, stable mixed chimerism, died 4 years after treatment from leukemia
Pulmonary embolus (Blood and lymphatic system disorders) | 1 (1) — Seven months after the transplant, one participant died from pulmonary embolus. Never developed GVHD
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hematopoietic Stem Cell Transplantation (N=4)
Step bovis infection (Infections and infestations) | 1 (1) — One participant had positive step bovis infection post-transplant. Pt had 2 previous step bovis infection prior to transplant. GI workup was negative and was cleared for transplant. The source for recurrent step bovis infection is unclear.
Urinary tract infection (UTI) (Infections and infestations) | 1 (1) — One participant had one episode of UTI treated with oral antibiotic
Sinus infection (Infections and infestations) | 1 (2) — One participant reported two sinus infections, one resolved without treatment, and one treated with oral antibiotic.

LIMITATIONS AND CAVEATS:
Small numbers of subjects enrolled

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes